CLINICAL TRIAL: NCT01771770
Title: Measurement of the Retinal Venous Pressure (RVP) Under Conditions of Chronically Reduced Ambient Pressure and Oxygen Partial Pressure (Field Study)
Brief Title: Measurement of Retinal Venous Pressure in Chronic Low-oxygen Environment
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: USB-2011-328
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: retinal venous pressure (RVP); chronically reduced ambient pressure; oxygen partial pressure; mountain sickness
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis is that the pressure in the retinal veins increases from chronic lack of oxygen and leads to decreased blood flow. On the basis of high altitude mountaineering this hypothesis should be verified. At the same time the adaptation capacity of the blood circulation should be analyzed, and a relationship to mountain sickness should be found.

DETAILED DESCRIPTION:
Conduct a field study to describe and quantify the retinal venous pressure (RVP) in healthy volunteers under conditions of controlled chronically reduced ambient pressure and oxygen partial pressure in the mountains. Obtaining indications regarding the adaptation of the retinal vascular system behavior to controlled, long-term hypoxic changes. Comparisons with blood pressure, pulse, oxygen saturation level and the appearance of symptoms of acute mountain sickness are made in order to obtain a better understanding of the development of high altitude illness.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* eye diseases
* systemic diseases
* term medication (except contraceptives)
* pregnancy
* allergies to the ingredients Alcain, Tropicamide and Phenylephrine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Quantify the changes in the retinal venous pressure (RVP). | 1-2 months
  Quantify the changes in the retinal venous pressure (RVP)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Flammer, MD, Study Director — University of Basel, Dept. of Ophthalmology
Locations (1):
- University of Basel, Dept. of Ophthalmology, Basel, Switzerland